CLINICAL TRIAL: NCT00155077
Title: The Correlation Between Tumor Angiogenesis and the Effect of Radiation Therapy in Cervical Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700771
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2004-06

CONDITIONS: Cervical Cancer
Keywords: cervical cancer, chemoradiotherapy, angiogenesis
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Carcinoma of the uterine cervix is a serious health problem. Cervical cancer is the most common malignant neoplasm of women in Taiwan. There were 2,720 new cases of invasive carcinoma of the cervix and 971 deaths from the disease in 2000. Cervical cancer is indeed is an important disease in Taiwan.

The primary therapies for cervical cancer are surgery, radiotherapy or chemoradiotherapy. Several clinical trials have showed that an improvement in time to progression and survival for patients given chemoradiotherapy compared with radiotherapy alone. Chemoradiotherapy is now regarded as standard modality to treat the locally advanced (stage IIB-IVA) or high-risk early-stage cervical cancer. However, some of the cervical cancer patients still failed to response to the treatment of cervical cancer or relapsed for completion of treatment.

Angiogenesis plays an important role in the pathogenesis of cancer. Recent studies have related angiogenesis to cancer growth and metastasis Ultrasonography has been used in the gynecologic field for decades. The previous studies of our team have shown that incremental angiogenesis could be demonstrated in the tumorigenesis of ovarian, endometrial malignancies, and cervical caner. Besides, other growth factors such as vascular endothelial growth factor (VEGF), and IL-6 have also been reported to correlate with the angiogenesis and the prognosis of cervical cancer. It seems that tumor angiogenesis could be utilized as a good marker to survey the severity of disease and prognosis of early-staged cervical cancer patients.

There is no good method or marker which could be utilized to monitor the response of radiotherapy and evaluate the prognosis of cervical cancer patients with advanced stages. So we would like to propose this proposal to focus on the tumor angiogenesis in cervical cancer patients with advanced stages. There are several purposes in this study. First, we will evaluate the kinetic changes of tumor angiogenesis in cervical cancer patients who receive radiotherapy or concurrent chemoradiotherapy. Second, we will evaluate that if the tumor angiogenesis could be a marker to monitor the response of radiotherapy or chemoradiotherapy in cervical cancer patients. The relation between tumor angiogenesis and radiotherapy will be explored and clarified by this study. The comprehensive role of tumor angiogenesis in cervical cancer will be elucidated by the results of this study.

DETAILED DESCRIPTION:
Carcinoma of the uterine cervix is a serious health problem. In Taiwan, cervical cancer is the most common malignant neoplasm and the 5th leading cause of cancer deaths in women (after carcinoma of the lung, liver, colorectum and breast). The Department of Health estimated that in 2000 there were 2,720 new cases of invasive carcinoma of the cervix and 971 deaths from the disease, in addition to more than 3,566 cases of carcinoma in situ (1).

The traditional treatment of invasive cervical cancer has been by surgery or radiotherapy or, certain situations, a combination of both. Most women with early-stage cervical cancers can be cured with radical surgery or radiotherapy. Those with a large cervical lesion at presentation or with spread to the pelvic lymph nodes or other pelvic tissues are usually treated with a combination of external-beam and intracavitary radiation. (2-6) To eradicate micrometastases and sensitize tumor cells to radiation, several studies have explored the use of radiotherapy with concomitant chemotherapy. (7-10) Because patients with cervical cancer usually present with disease that is clinically confined to the pelvis, locoregional disease control is the primary challenge for physicians. Treatment with carefully tailored surgery or radiotherapy has produced impressive cure rates in patients with early-stage disease. Primary radiotherapy for early-stage disease offers cure rates equivalent to those with radical hysterectomy. For more locally advanced disease, with spread beyond the uterus (stage IIB to IVA according to the staging system of the International Federation of Gynecology and Obstetrics), radiotherapy is the primary modality of treatment. For these patients, cure rates decrease with advancing stage and tumor bulk. (11) A significant reason for treatment failure in many patients is the inability to achieve control over the primary cancer and first-echelon lymph node metastases. (12) Improvement in local control can be expected to lead to improved cure rates. (13) Simply increasing the dose of RT will increase local control rates, but it does so at the expense of increased complication rates. (14) Once cervical cancer has extended beyond the cervix, cure with radical surgery alone is unlikely. After reports from several randomized clinical trials showing an improvement in time to progression and survival for patients given chemoradiotherapy compared with radiotherapy alone. (15-18) the chemoradiotherapy should be considered as standard care for locally advanced (stage IIB-IVA) or high-risk early-stage cervical cancer.

Radical radiotherapy is effective for patients with locoregionally confined cervical cancer of any stage. Treatment must be carefully tailored to the patient and to the extent of disease but usually consists of a combination of external-beam irradiation and brachytherapy. Overall, reported 5-year survival rates of patients treated with radiation alone are approximately 75% to 85% for stage IB , 65% to 75% for stage II, 30% to 50% for stage III, and 10% to 20% for stage IVA disease. Within stage subsets, cure rates are strongly correlated with the size of the primary tumor and the extent of regional involvement.(17, 18) For locally advanced disease, a systematic review and meta-analysis of reports on the use of chemoradiotherapy generally supported the use of chemoradiotherapy over radiotherapy alone, or neoadjuvant chemotherapy followed by radiotherapy. (19) Chemoradiotherapy showed to improve overall survival by about 30% and reduced the risk of both local and distant recurrence. Absolute survival benefit was estimated as 12%, though several studies have reported higher survival benefits.

Angiogenesis plays an important role in the pathogenesis of cancer (20). Recent studies have related angiogenesis to cancer growth and metastasis(21). The growth of solid tumors and their metastatic spread is angiogenesis dependent and this has been confirmed in several experimental and clinical studies (22, 23). Ultrasonography has been used in the gynecologic field for decades. Our previous studies have shown that incremental angiogenesis could be demonstrated in the tumorigenesis of ovarian, endometrial malignancies, and cervical caner. (24-28) Besides, other growth factors such as vascular endothelial growth factor (VEGF), and IL-6 have also been reported to correlate with the angiogenesis and the prognosis of cervical cancer (29-31), ovarian cancer (32), and endometrial cancer (27, 33). Tumor angiogenesis of cervical cancer has been proved to be correlated with the disease severity and prognosis of the cervical cancer patients with early stages (26, 29, 30, 34). It seems that tumor angiogenesis could be utilized as a good marker to survey the severity of disease and prognosis of early-staged cervical cancer patients.

However, there is no good method or marker which could be utilized to monitor the response of radiotherapy and evaluate the prognosis of cervical cancer patients with advanced stages. So we would like to propose this proposal to focus on the tumor angiogenesis in cervical cancer patients with advanced stages. Cervical cancer patients who will receive radiotherapy or concurrent chemoradiotherapy will be enrolled in this study. Transvaginal sonography and angiogenesis-related growth factors will be evaluated to monitor and response of treatment in each patient. There are several purposes in this study. First, we will evaluate the kinetic changes of tumor angiogenesis in cervical cancer patients who receive radiotherapy or concurrent chemoradiotherapy. Second, we will evaluate that if the tumor angiogenesis could be a marker to monitor the response of radiotherapy or concurrent chemoradiotherapy in cervical cancer patients. The relation between tumor angiogenesis and radiotherapy will be explored and clarified by this study. The comprehensive role of tumor angiogenesis in cervical cancer will be elucidated by the results of this study.

ELIGIBILITY:
Inclusion Criteria:

- cervical cancer patients receiving radiotherapy or chemo-radiotherapy

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-06; Study Completion 2009-06

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yuan Huang, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan